CLINICAL TRIAL: NCT06197074
Title: Evaluation of Morphologic Parameters of Quadriceps Muscle Predicting Disease Activity, Physical Performance and Quality of Life in Women With Rheumatoid Arthritis
Brief Title: Effect of Quadriceps Muscle on Physical Outcome Measures in Women With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Erdal Horata, PhD; Lecturer; Principal Investigator, Afyonkarahisar Health Sciences University
Other Study IDs: 2023/8
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasound assessment — The morphological characteristics of the quadriceps muscle of the participants will be assessed using ultrasound.

SUMMARY:
Studies have reported that individuals with Rheumatoid Arthritis have a smaller muscle cross-sectional area, pennation angle and muscle thickness than healthy controls. Sarcopenia may decrease physical performance and quality of life in individuals with RA. Therefore, morphologic changes in the quadriceps femoris muscle due to sarcopenia may help us to gain insight into physical function and quality of life. This study aims to evaluate the predictive capacity of morphologic characteristics of the quadriceps femoris muscle for disease activity, physical performance, and quality of life in women with Rheumatoid Arthritis.

DETAILED DESCRIPTION:
Studies have reported that individuals with Rheumatoid Arthritis have a smaller muscle cross-sectional area, pennation angle and muscle thickness than healthy controls. Sarcopenia may decrease physical performance and quality of life in individuals with RA. Therefore, morphologic changes in the quadriceps femoris muscle due to sarcopenia may help us to gain insight into physical function and quality of life. This study aims to evaluate the predictive capacity of morphologic characteristics of the quadriceps femoris muscle for disease activity, physical performance, and quality of life in women with Rheumatoid Arthritis.

Within the scope of the study, the morphological characteristics of the quadriceps muscle of the participants will be evaluated by a Physical Medicine and Rehabilitation specialist physician via ultrasound. After appropriate visualization, the image will be captured and saved in JPEG format, and will be exported to the ImageJ program for further analysis and evaluations will be performed by an anatomist. Assessments of quality of life and physical performance will be made by a physiotherapist involved in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* Female participants with a confirmed diagnosis of RA for at least 3 years according to the 2010 American College of Rheumatology (ACR) criteria
* Presence of sarcopenia

Exclusion Criteria:

* Presence of fractures, burns or lesions in the area to be measured
* Presence of any neuromuscular, cardiovascular or metabolic disease,
* Individuals with knee endoprosthesis,
* Inability to walk

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female participants between the ages of 18-65 who have been diagnosed with Rheumatoid Arthritis for at least 3 years and who come to Afyonkarahisar Health Sciences University Physical Therapy and Rehabilitation outpatient clinic will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Vastus lateralis muscle length | 10 minutes
  Vastus Lateralis muscle length will be measured bilaterally by Ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: ERDAL HORATA, PhD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided